CLINICAL TRIAL: NCT00984620
Title: Antiviral Effect and Safety of Once Daily BI 201335 NA in Hepatitis C Virus Genotype 1 Infected Treatment-naive Patients for 12 or 24 Weeks as Combination Therapy With Pegylated Interferon-alpha 2a and Ribavirin (Randomised, Open Label, Phase II)
Brief Title: Short Term Treatment With BI 201335, Peginterferon-alpha 2a and Ribavirin in Hepatitis c Virus Genotype-1 Treatment-naïve Patients (SILEN-C3)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1220.40; 2009-012579-90 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — faldaprevir; Ribavirin

ARMS (2):
- short arm (Experimental): patients to receive BI201335 with PegIFN/RBV for 12 wks followed by 12 weeks PegIFN/RBV with a 3 days lead-in phase of PegIFN/RBV (i.e. initiation of BI 201335 NA 3 days after first administration of PegIFN/RBV)
  Interventions: Drug: BI 201335; Drug: Pegylated Interferon-alpha (IFN); Drug: Ribavirin (RBV)
- long arm (Experimental): patients to receive BI201335 with PegIFN/RBV for 24 wks with a 3 days lead-in phase of PegIFN/RBV (i.e. initiation of BI 201335 NA 3 days after first administration of PegIFN/RBV)
  Interventions: Drug: BI 201335; Drug: Pegylated Interferon-alpha (IFN); Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: BI 201335 — BI 201335
  Arms: long arm
Drug: BI 201335 — BI 201335
  Arms: short arm
Drug: Pegylated Interferon-alpha (IFN) — Pegylated Interferon-alpha
Drug: Ribavirin (RBV) — Ribavirin (RBV)

SUMMARY:
To compare the antiviral efficacy and safety of a 12-week with a 24-week treatment of BI 201335 at a dose of 120 mg once daily, with a 24-week background of pegylated interferon-alpha 2a (PegIFN) plus ribavirin (RBV), in treatment-naïve patients infected with hepatitis C virus (HCV) genotype 1

ELIGIBILITY:
Inclusion criteria:

1. Chronic hepatitis C infection of genotype 1
2. Therapy-naïve to interferon, pegylated interferon, and ribavirin
3. HCV viral load > 100.000 IU/ml at screening
4. Liver biopsy or fibroscan within two years prior to screening that provides evidence of any degree of fibrosis or cirrhosis
5. Normal retinal finding on fundoscopy within 6 months prior to Day 1
6. Age 18 to 70 years

Exclusion criteria:

1. HCV of mixed genotype (1/2, 1/3, and 1/4) .
2. Patients who have been previously treated with at least one dose of any protease inhibitor
3. Evidence of liver disease due to causes other than chronic HCV infection
4. Positive for HIV-1 or HIV-2 antibodies
5. Hepatitis B virus (HBV) infection
6. Decompensated liver disease, or history of decompensated liver disease
7. Active malignancy or history of malignancy within the last 5 years
8. History of alcohol or drug abuse (except cannabis) within the past 12 months.
9. Body Mass Index < 18 or > 35 kg/m2.
10. Usage of any investigational drugs within 30 days prior to enrolment
11. Alpha fetoprotein value >100ng/mL at screening;
12. Total bilirubin > 1.5 x ULN with ratio of direct/indirect > 1.
13. ALT or AST level > 10 x ULN

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (28):
- United States (6):
  - 1220.40.002 Boehringer Ingelheim Investigational Site, Tulepo, Mississippi
  - 1220.40.007 Boehringer Ingelheim Investigational Site, New York, New York
  - 1220.40.006 Boehringer Ingelheim Investigational Site, Germantown, Tennessee
  - 1220.40.004 Boehringer Ingelheim Investigational Site, Jackson, Tennessee
  - 1220.40.003 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 1220.40.005 Boehringer Ingelheim Investigational Site, Austin, Texas
- Austria (2):
  - 1220.40.4303 Boehringer Ingelheim Investigational Site, Linz
  - 1220.40.4301 Boehringer Ingelheim Investigational Site, Vienna
- Canada (5):
  - 1220.40.1004 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1220.40.1001 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1220.40.1002 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1220.40.1003 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1220.40.1005 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- France (6):
  - 1220.40.3303A Boehringer Ingelheim Investigational Site, Clichy
  - 1220.40.3305A Boehringer Ingelheim Investigational Site, Lille
  - 1220.40.3301A Boehringer Ingelheim Investigational Site, Marseille
  - 1220.40.3306A Boehringer Ingelheim Investigational Site, Montpellier
  - 1220.40.3302A Boehringer Ingelheim Investigational Site, Paris
  - 1220.40.3304A Boehringer Ingelheim Investigational Site, Rennes
- Germany (6):
  - 1220.40.4902 Boehringer Ingelheim Investigational Site, Berlin
  - 1220.40.4909 Boehringer Ingelheim Investigational Site, Berlin
  - 1220.40.4906 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1220.40.4908 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1220.40.4904 Boehringer Ingelheim Investigational Site, Hamburg
  - 1220.40.4905 Boehringer Ingelheim Investigational Site, Mainz
- Romania (3):
  - 1220.40.4001 Boehringer Ingelheim Investigational Site, Bucharest
  - 1220.40.4002 Boehringer Ingelheim Investigational Site, Bucharest
  - 1220.40.4003 Boehringer Ingelheim Investigational Site, Bucharest

REFERENCES:
- [Derived] Dieterich D, Asselah T, Guyader D, Berg T, Schuchmann M, Mauss S, Ratziu V, Ferenci P, Larrey D, Maieron A, Stern JO, Ozan M, Datsenko Y, Bocher WO, Steinmann G. SILEN-C3, a phase 2 randomized trial with faldaprevir plus pegylated interferon alpha-2a and ribavirin in treatment-naive hepatitis C virus genotype 1-infected patients. Antimicrob Agents Chemother. 2014 Jun;58(6):3429-36. doi: 10.1128/AAC.02497-13. Epub 2014 Apr 7. PMID 24709256

RESULTS

PARTICIPANT FLOW:
Groups:
- Faldaprevir 120mg (12 Weeks): Patients received Faldaprevir (BI201335) 120 mg soft gelatine capsule once daily combined with PegIFN/RBV (Pegylated interferon alpha-2a solution for injection/Ribavirin tablet) for 12 weeks, with a 3 days lead-in phase of PegIFN/RBV (i.e. initiation of Faldaprevir (BI201335) 3 days after first administration of PegIFN/RBV), followed by PegIFN/RBV for additional 12 weeks. Patients who did not show an extended early virological response (eRVR) continued treatment with PegIFN/RBV alone for a total of 24 to 48 weeks.
- Faldaprevir 120mg (24 Weeks): Patients received Faldaprevir (BI201335) 120 mg soft gelatine capsule once daily combined with PegIFN/RBV (Pegylated interferon alpha-2a solution for injection/Ribavirin tablet) for 24 weeks, with a 3 days lead-in phase of PegIFN/RBV (i.e. initiation of Faldaprevir (BI201335) 3 days after first administration of PegIFN/RBV). Patients who did not show an extended early virological response (eRVR) continued treatment with PegIFN/RBV alone for a total of 24 to 48 weeks.
Period: Overall Study
Arm/Group | Faldaprevir 120mg (12 Weeks) | Faldaprevir 120mg (24 Weeks)
Started | 81 | 79
Completed | 75 | 67
Not Completed | 6 | 12
Not completed — Adverse Event | 5 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — reason other than listed above | 0 | 4

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): contained all randomised patients who were dispensed study medication and were documented to have taken at least one dose of study medication.
Groups:
- Faldaprevir 120 mg (12 Weeks): Patients received Faldaprevir (BI201335) 120 mg soft gelatine capsule once daily combined with PegIFN/RBV (Pegylated interferon alpha-2a solution for injection/Ribavirin tablet) for 12 weeks, with a 3 days lead-in phase of PegIFN/RBV (i.e. initiation of Faldaprevir (BI201335) 3 days after first administration of PegIFN/RBV), followed by PegIFN/RBV for additional 12 weeks. Patients who did not show an extended early virological response (eRVR) continued treatment with PegIFN/RBV alone for a total of 24 to 48 weeks.
- Faldaprevir 120 mg (24 Weeks): Patients received Faldaprevir (BI201335) 120 mg soft gelatine capsule once daily combined with PegIFN/RBV (Pegylated interferon alpha-2a solution for injection/Ribavirin tablet) for 24 weeks, with a 3 days lead-in phase of PegIFN/RBV (i.e. initiation of Faldaprevir (BI201335) 3 days after first administration of PegIFN/RBV). Patients who did not show an extended early virological response (eRVR) continued treatment with PegIFN/RBV alone for a total of 24 to 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Faldaprevir 120 mg (12 Weeks) | Faldaprevir 120 mg (24 Weeks) | Total
Number analyzed (Participants) | 81 | 79 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (9.4) | 44.9 (11.9) | 46.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 34 | 61
  Male | 54 | 45 | 99

OUTCOME MEASURES:

1. Primary Outcome: Virological Response at Week 28 (W28VR)
Description: Virological response at Week 28: The patients who reached plasma hepatitis C virus ribonucleic acid (HCV RNA) level below the lower limit of detection (BLD) at Week 28.
Time Frame: 28 weeks
Population: Per Protocol Set (PPS): included all patients in the FAS without important protocol deviations.
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120 mg (12 Weeks) | Faldaprevir 120 mg (24 Weeks)
Number analyzed (Participants) | 81 | 78
participants | 61 | 60
Statistical Analysis 1: Comparison: Faldaprevir 120 mg (12 Weeks) vs Faldaprevir 120 mg (24 Weeks); Test type: Superiority or Other; p = 0.855, Cochran-Mantel-Haenszel; Based on an Cochran-Mantel-Haenszel method adjusted by HCV genotype (1a and 1b only); Adjusted percent difference = -1.25, 95% CI 2-sided [-14.3 to 11.8] — p-value presented is 2-sided. The percent differences and p-values are based on a comparison to the Faldaprevir 120mg (12 Weeks)

2. Secondary Outcome: Rapid Virological Response at Week 4 (RVR)
Description: Rapid virological response at week 4 (RVR): The patients who reached plasma hepatitis C virus ribonucleic acid (HCV RNA) level below the lower limit of detection (BLD) at week 4.
Time Frame: 4 weeks
Population: PPS
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120 mg (12 Weeks) | Faldaprevir 120 mg (24 Weeks)
Number analyzed (Participants) | 81 | 78
participants | 48 | 56
Statistical Analysis 1: Comparison: Faldaprevir 120 mg (12 Weeks) vs Faldaprevir 120 mg (24 Weeks); Test type: Superiority or Other; p = 0.229, Cochran-Mantel-Haenszel; Based on an Cochran-Mantel-Haenszel method adjusted by HCV genotype (1a and 1b only); Adjusted percent difference = 9.02, 95% CI 2-sided [-5.3 to 23.3] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Virological Response at Week 24 (W24VR)
Description: virological response at week 24 (W24VR): The patients who reached plasma hepatitis C virus ribonucleic acid (HCV RNA) level below the lower limit of detection (BLD) at week 24.
Time Frame: 24 weeks
Population: PPS
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120 mg (12 Weeks) | Faldaprevir 120 mg (24 Weeks)
Number analyzed (Participants) | 81 | 78
participants | 59 | 63
Statistical Analysis 1: Comparison: Faldaprevir 120 mg (12 Weeks) vs Faldaprevir 120 mg (24 Weeks); Test type: Superiority or Other; p = 0.417, Cochran-Mantel-Haenszel; Based on an Cochran-Mantel-Haenszel method adjusted by HCV genotype (1a and 1b only); Adjusted percent difference = 5.48, 95% CI 2-sided [-7.3 to 18.3] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Virological Response at Week 36 (W36VR)
Description: Virological response at week 36 (W36VR): the patients who reached plasma hepatitis C virus ribonucleic acid (HCV RNA) level below the lower limit of detection (BLD) at week 36.
Time Frame: 36 weeks
Population: PPS
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120 mg (12 Weeks) | Faldaprevir 120 mg (24 Weeks)
Number analyzed (Participants) | 81 | 78
participants | 55 | 58
Statistical Analysis 1: Comparison: Faldaprevir 120 mg (12 Weeks) vs Faldaprevir 120 mg (24 Weeks); Test type: Superiority or Other; p = 0.676, Cochran-Mantel-Haenszel; Based on an Cochran-Mantel-Haenszel method adjusted by HCV genotype (1a and 1b only); Adjusted percent difference = 2.99, 95% CI 2-sided [-10.6 to 16.6] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: End of Treatment Response (ETR)
Description: End of Treatment Response (ETR): The patients who reached plasma hepatitis C virus ribonucleic acid (HCV RNA) level below the lower limit of detection (BLD) at end of all therapy.
Time Frame: up to 48 weeks
Population: PPS
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120 mg (12 Weeks) | Faldaprevir 120 mg (24 Weeks)
Number analyzed (Participants) | 81 | 78
participants | 65 | 67
Statistical Analysis 1: Comparison: Faldaprevir 120 mg (12 Weeks) vs Faldaprevir 120 mg (24 Weeks); Test type: Superiority or Other; p = 0.588, Cochran-Mantel-Haenszel; Based on an Cochran-Mantel-Haenszel method adjusted by HCV genotype (1a and 1b only); Adjusted percent difference = 3.24, 95% CI 2-sided [-8.1 to 14.6] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Sustained Virological Response (SVR24) at 24 Weeks After Completion of All Therapy
Description: Sustained Virological Response (SVR24) at 24 weeks: The patients who reached plasma Hepatitis C virus Ribonucleic acid (HCV RNA) level below the lower limit of detection (BLD) at 24 weeks after completion of all Hepatitis C virus (HCV) therapy.
Time Frame: 72 weeks
Population: PPS
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120 mg (12 Weeks) | Faldaprevir 120 mg (24 Weeks)
Number analyzed (Participants) | 81 | 78
participants | 54 | 58
Statistical Analysis 1: Comparison: Faldaprevir 120 mg (12 Weeks) vs Faldaprevir 120 mg (24 Weeks); Test type: Superiority or Other; p = 0.512, Cochran-Mantel-Haenszel; Based on an Cochran-Mantel-Haenszel method adjusted by HCV genotype (1a and 1b only); Adjusted percent difference = 4.78, 95% CI 2-sided [-9.0 to 18.6] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Viral Load (HCV RNA) at All Visits During Treatment and Follow-up
Description: Viral load of Hepatitis C virus Ribonucleic acid (HCV RNA) at all visits during treatment (TRT) and follow-up, ie. change from baseline viral load at all visits.
Time Frame: From baseline to 72 weeks
Population: PPS
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Faldaprevir 120 mg (12 Weeks) | Faldaprevir 120 mg (24 Weeks)
Number analyzed (Participants) | 81 | 78
IU/mL
  week 2, change from baseline (N=76, N=78) | -4.724 (0.9059) | -4.866 (0.8664)
  week 4, change from baseline (N=76, N=77) | -4.993 (1.1168) | -5.081 (1.1195)
  week 8, change from baseline (N=75, N=76) | -5.128 (1.1159) | -5.088 (1.3150)
  week 12, change from baseline (N=76, N=76) | -5.117 (1.1495) | -5.107 (1.2852)
  week 16, change from baseline (N=18, N=13) | -5.363 (1.2341) | -5.262 (0.5820)
  week 20, change from baseline (N=52, N=57) | -5.056 (1.0894) | -5.366 (0.7319)
  week 24, change from baseline (N=12, N=8) | -4.176 (2.1635) | -4.740 (1.6576)
  week 28, change from baseline (N=4, N=4) | -5.723 (0.6795) | -4.369 (2.2917)
  week 36, change from baseline (N=4, N=2) | -5.624 (0.7059) | -5.958 (0.1909)
  End of TRT, change from baseline (N=80, N=78) | -4.910 (1.4690) | -5.017 (1.4434)
  4 wks after TRT, change from baseline (N=75, N=77) | -4.296 (2.2499) | -4.367 (2.1849)
  12 wks after TRT, change from baseline (N=75,N=75) | -4.154 (2.3356) | -4.353 (2.1588)
  24 wks after TRT, change from baseline (N=73,N=75) | -4.103 (2.3673) | -4.250 (2.2439)

8. Secondary Outcome: Time to Reach a Plasma HCV RNA Level BLD While on Treatment
Description: Time to reach a plasma Hepatitis C Virus Ribonucleic Acid (HCV RNA) level below the lower limit of detection (BLD) while on treatment
Time Frame: 48 weeks
Population: PPS
Measure: Median (Inter-Quartile Range); unit: week
Arm/Group | Faldaprevir 120 mg (12 Weeks) | Faldaprevir 120 mg (24 Weeks)
Number analyzed (Participants) | 81 | 78
week | 4.1 [4 to 8] | 4.1 [2 to 8]
Statistical Analysis 1: Comparison: Faldaprevir 120 mg (12 Weeks) vs Faldaprevir 120 mg (24 Weeks); Test type: Superiority or Other; p = 0.1397, Log Rank — Compare 120 MG Faldaprevir 120mg (24 Weeks) over 120 MG Faldaprevir 120mg (12 Weeks) using log-rank test

9. Secondary Outcome: Laboratory Test Abnormalities and Study Medication Tolerabilities
Description: Participants with possible clinically significant laboratory test abnormalities observed in functional groups: Haematology, Coagulation, Electrolytes, Enzymes, Substrates and Differentials, automatic.
Time Frame: 48 weeks
Population: Treated Set (TS): comprised all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment regardless of randomisation.
Measure: Number; unit: participants
Arm/Group | Faldaprevir 120 mg (12 Weeks) | Faldaprevir 120 mg (24 Weeks)
Number analyzed (Participants) | 81 | 79
participants
  Red blood cell count: low (N=81, N=79) | 9 | 8
  haematocrit: low (N=81, N=79) | 30 | 21
  haematocrit: high(N=81, N=79) | 0 | 1
  white blood cell count: low(N=81, N=79) | 56 | 60
  platelets: low(N=81, N=78) | 5 | 2
  eosinophils: high (N=81, N=79) | 1 | 5
  PT-INR: high (N=81, N=79) | 1 | 1
  sodium: low (N=81, N=79) | 1 | 1
  bicarbonate: low (N=79, N=74) | 6 | 11
  bicarbonate: high (N=79, N=74) | 1 | 1
  AST/GOT, SGOT: high (N=75, N=71) | 3 | 3
  ALT/GPT, SGPT: high (N=68, N=64) | 3 | 5
  alkaline phosphatase: high (N=80, N=79) | 1 | 0
  GGT: high (N=74, N=72) | 4 | 8
  creatine kinase: high (N=80, N=79) | 0 | 3
  lipase: high (N=79, N=79) | 1 | 3
  amylase: high (N=81, N=79) | 1 | 2
  glucose: low (N=80, N=79) | 0 | 2
  cholesterol, total: high (N=80, N=75) | 6 | 2
  triglyceride: high (N=74, N=71) | 13 | 18

10. Secondary Outcome: Number of Participants With Clinically Relevant Abnormalities Vital Signs, and Physical Examination
Description: No number of participants with clinically relevant abnormalities in vital signs and physical examination.
Time Frame: 48 weeks
Population: TS
Measure: Number; unit: participants with abnormality
Arm/Group | Faldaprevir 120mg (12 Weeks) | Faldaprevir 120mg (24 Weeks)
Number analyzed (Participants) | 81 | 79
participants with abnormality | 0 | 0

11. Secondary Outcome: Laboratory Test Value Changes Over Time for Selected Lab Test Parameters (1)
Description: Change from baseline (CFB) in Red blood cells.
Time Frame: baseline and 48 weeks
Population: TS
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Faldaprevir 120mg (12 Weeks) | Faldaprevir 120mg (24 Weeks)
Number analyzed (Participants) | 81 | 79
10^12 cells/L
  Red blood cell (10^12cells/L) CFB,Day 1(N=77,N=75) | 0.0 (0.3) | -0.1 (0.3)
  Red blood cell (10^12cells/L) CFB, wk2 (N=75,N=77) | -0.3 (0.5) | -0.4 (0.5)
  Red blood cell (10^12cells/L) CFB, wk4(N=74, N=76) | -0.8 (0.5) | -0.8 (0.6)
  Red blood cell (10^12cells/L) CFB, wk8(N=75, N=74) | -1.0 (0.5) | -1.0 (0.5)
  Red blood cell (10^12cells/L) CFB, wk12(N=74,N=74) | -1.1 (0.6) | -1.2 (0.5)
  Red blood cell (10^12cells/L) CFB, wk18(N=66,N=69) | -1.2 (0.6) | -1.2 (0.5)
  Red blood cell (10^12cells/L) CFB, wk24(N=12, N=4) | -1.2 (0.7) | -0.9 (0.4)
  Red blood cell (10^12cells/L) CFB, wk28(N=4, N=3) | -1.1 (0.4) | -0.9 (0.7)
  Red blood cell (10^12cells/L) CFB, wk36(N=4, N=2) | -0.9 (0.9) | -1.4 (0.2)
  Red blood cell (10^12cells/L) CFB, EoT(N=67, N=73) | -1.2 (0.6) | -1.2 (0.5)

12. Secondary Outcome: Laboratory Test Value Changes Over Time for Selected Lab Test Parameters (2)
Description: Change from baseline (CFB) in haematocrit and Eosinophils.
Time Frame: baseline and 48 weeks
Population: TS
Measure: Mean (Standard Deviation); unit: % of laboratory test substance
Arm/Group | Faldaprevir 120mg (12 Weeks) | Faldaprevir 120mg (24 Weeks)
Number analyzed (Participants) | 81 | 79
% of laboratory test substance
  haematocrit (%) CFB, Day1 (N=77, N=75) | -0.9 (3.0) | -1.3 (2.7)
  haematocrit (%) CFB, wk2 (N=75, N=77) | -4.3 (4.4) | -4.7 (4.2)
  haematocrit (%) CFB, wk4 (N=74, N=76) | -8.0 (4.9) | -7.9 (4.5)
  haematocrit (%) CFB, wk8 (N=75, N=74) | -8.4 (4.6) | -7.1 (4.0)
  haematocrit (%) CFB, wk12 (N=72, N=74) | -8.5 (4.9) | -7.8 (3.9)
  haematocrit (%) CFB, wk18 (N=66, N=69) | -7.3 (5.4) | -6.5 (4.4)
  haematocrit (%) CFB, wk24 (N=11, N=4) | -6.6 (6.2) | -2.7 (2.4)
  haematocrit (%) CFB, wk28 (N=4, N=3) | -3.8 (3.9) | -1.2 (4.4)
  haematocrit (%) CFB, wk36 (N=4, N=2) | -3.0 (8.0) | -3.6 (0.0)
  haematocrit (%) CFB, EoT (N=66, N=70) | -6.0 (4.7) | -6.0 (4.6)
  Eosinophils(%), CFB, day1 (N=77, N=75) | 0 (1) | 0 (1)
  Eosinophils(%), CFB, wk2 (N=75, N=76) | 0 (2) | 0 (1)
  Eosinophils(%), CFB, wk4 (N=73, N=74) | -1 (1) | 0 (2)
  Eosinophils(%), CFB, wk8 (N=74, N=73) | 0 (2) | 0 (5)
  Eosinophils(%), CFB, wk12 (N=72, N=72) | 0 (2) | 0 (3)
  Eosinophils(%), CFB, wk18 (N=62, N=65) | 0 (3) | 0 (2)
  Eosinophils(%), CFB, wk24 (N=12, N=4) | -1 (1) | -1 (2)
  Eosinophils(%), CFB, wk28 (N=4, N=3) | -1 (1) | -2 (2)
  Eosinophils(%), CFB, wk36 (N=4, N=2) | -1 (1) | -1 (0)
  Eosinophils(%), CFB, EoT (N=66, N=70) | 0 (2) | 1 (5)

13. Secondary Outcome: Laboratory Test Value Changes Over Time for Selected Lab Test Parameters (3)
Description: Change from baseline (CFB) in Platelets and white blood cells.
Time Frame: baseline and 48 weeks
Population: TS
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Faldaprevir 120mg (12 Weeks) | Faldaprevir 120mg (24 Weeks)
Number analyzed (Participants) | 81 | 79
10^9 cells/L
  Platelets CFB, Day 1 (N=77, N=73) | 3 (35) | 2 (29)
  Platelets CFB, wk2 (N=74, N=74) | -35 (40) | -35 (34)
  Platelets CFB, wk4 (N=73, N=74) | -35 (41) | -39 (42)
  Platelets CFB, wk8 (N=73, N=71) | -55 (37) | -48 (38)
  Platelets CFB, wk12 (N=72, N=72) | -61 (38) | -50 (40)
  Platelets CFB, wk18 (N=66, N=68) | -55 (46) | -51 (45)
  Platelets CFB, wk24 (N=12, N=3) | -46 (37) | -50 (43)
  Platelets CFB, wk28 (N=4, N=2) | -22 (77) | -83 (6)
  Platelets CFB, wk36 (N=4, N=2) | -47 (31) | -85 (2)
  Platelets CFB, EoT (N=67, N=71) | -59 (46) | -50 (48)
  white blood cell CFB, day1 (N=77, N=75) | -0.1 (1.1) | 0.3 (1.3)
  white blood cell CFB, wk2 (N=75, N=77) | -2.2 (1.5) | -1.8 (1.9)
  white blood cell CFB, wk4 (N=74, N=76) | -2.6 (1.5) | -2.6 (1.9)
  white blood cell CFB, wk8 (N=75, N=74) | -3.2 (1.5) | -2.9 (1.4)
  white blood cell CFB, wk12 (N=74, N=74) | -3.4 (1.5) | -2.8 (1.8)
  white blood cell CFB, wk18 (N=66, N=69) | -3.2 (1.4) | -3.1 (1.6)
  white blood cell CFB, wk24 (N=12, N=4) | -4.0 (1.3) | -2.0 (1.7)
  white blood cell CFB, wk28 (N=4, N=3) | -2.8 (1.0) | -1.9 (2.0)
  white blood cell CFB, wk36 (N=4, N=2) | -2.5 (0.9) | -3.0 (1.1)
  white blood cell CFB, EoT (N=67, N=73) | -3.4 (1.5) | -3.1 (1.6)

14. Secondary Outcome: Laboratory Test Value Changes Over Time for Selected Lab Test Parameters (4)
Description: Change from baseline (CFB) in Sodium, Bicarbonate, Cholesterol total, Triglyceride, and Glucose.
Time Frame: baseline and 48 weeks
Population: TS
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faldaprevir 120mg (12 Weeks) | Faldaprevir 120mg (24 Weeks)
Number analyzed (Participants) | 81 | 79
mmol/L
  Sodium (mmol/L) CFB, Day 1(N=77, N=74) | 0 (2) | 1 (2)
  Sodium (mmol/L) CFB, wk2 (N=76, N=78) | 0 (2) | 0 (2)
  Sodium (mmol/L) CFB, wk4 (N=76, N=77) | 0 (2) | 0 (2)
  Sodium (mmol/L) CFB, wk8 (N=73, N=76) | 1 (3) | 1 (2)
  Sodium (mmol/L) CFB, wk12 (N=75, N=76) | 0 (2) | 1 (2)
  Sodium (mmol/L) CFB, wk18 (N=68, N=70) | 0 (2) | 0 (2)
  Sodium (mmol/L) CFB, wk24 (N=12, N=4) | -1 (2) | 0 (1)
  Sodium (mmol/L) CFB, wk28 (N=5, N=3) | -2 (2) | -1 (3)
  Sodium (mmol/L) CFB, wk36 (N=4, N=2) | -1 (2) | -1 (2)
  Sodium (mmol/L) CFB, EoT (N=67, N=73) | 0 (2) | 0 (3)
  Bicarbonate (mmol/L), CFB, day1 (N=76, N=75) | 0.1 (1.4) | 0.2 (1.3)
  Bicarbonate (mmol/L), CFB, wk2 (N=75, N=78) | -0.2 (1.4) | 0.0 (1.3)
  Bicarbonate (mmol/L), CFB, wk4 (N=74, N=77) | -0.1 (1.3) | -0.1 (1.3)
  Bicarbonate (mmol/L), CFB, wk8 (N=74, N=76) | -0.1 (1.3) | 0.0 (1.4)
  Bicarbonate (mmol/L), CFB, wk12 (N=74, N=76) | -0.3 (1.2) | -0.4 (1.5)
  Bicarbonate (mmol/L), CFB, wk18 (N=66, N=69) | -0.3 (1.6) | -0.4 (1.3)
  Bicarbonate (mmol/L), CFB, wk24 (N=12, N=4) | -0.4 (1.4) | -0.5 (1.9)
  Bicarbonate (mmol/L), CFB, wk28 (N=4, N=3) | -1.2 (2.1) | -0.2 (0.9)
  Bicarbonate (mmol/L), CFB, wk36 (N=4, N=2) | -2.6 (2.3) | -1.0 (0.7)
  Bicarbonate (mmol/L), CFB, EoT (N=64, N=71) | -0.2 (1.6) | -0.1 (1.4)
  Cholesterol tot. (mmol/L), CFB, day1 (n=77, N=75) | 0.03 (0.47) | -0.05 (0.48)
  Cholesterol tot. (mmol/L), CFB, wk2 (n=76, N=78) | -0.48 (0.57) | -0.54 (0.57)
  Cholesterol tot. (mmol/L), CFB, wk4 (n=76, N=77) | -0.51 (0.55) | -0.67 (0.68)
  Cholesterol tot. (mmol/L), CFB, wk8 (n=75, N=76) | -0.58 (0.59) | -0.60 (0.62)
  Cholesterol tot. (mmol/L), CFB, wk12 (n=75, N=76) | -0.64 (0.62) | -0.74 (0.63)
  Cholesterol tot. (mmol/L), CFB, wk18 (n=68, N=70) | -0.51 (0.64) | -0.80 (0.69)
  Cholesterol tot. (mmol/L), CFB, wk24 (n=12, N=4) | -0.36 (0.46) | -0.37 (0.30)
  Cholesterol tot. (mmol/L), CFB, wk28 (n=5, N=3) | 0.10 (0.53) | -0.09 (0.20)
  Cholesterol tot. (mmol/L), CFB, wk36 (n=4, N=2) | -0.35 (0.14) | -0.23 (0.20)
  Cholesterol tot. (mmol/L), CFB, EoT (n=67, N=73) | -0.43 (0.70) | -0.74 (0.68)
  Triglyceride (mmol/L), CFB, day1 (N=77, N=75) | -0.1 (0.5) | -0.1 (0.3)
  Triglyceride (mmol/L), CFB, wk2 (N=76, N=78) | 0.1 (0.5) | 0.1 (0.4)
  Triglyceride (mmol/L), CFB, wk4 (N=76, N=77) | 0.1 (0.5) | 0.2 (0.6)
  Triglyceride (mmol/L), CFB, wk8 (N=75, N=76) | 0.1 (0.5) | 0.1 (0.4)
  Triglyceride (mmol/L), CFB, wk12 (N=75, N=76) | 0.1 (0.6) | 0.1 (0.5)
  Triglyceride (mmol/L), CFB, wk18 (N=68, N=70) | 0.0 (0.5) | 0.2 (0.5)
  Triglyceride (mmol/L), CFB, wk24 (N=12, N=4) | -0.2 (0.7) | 0.2 (0.3)
  Triglyceride (mmol/L), CFB, wk28 (N=5, N=3) | 0.0 (1.3) | 0.4 (0.4)
  Triglyceride (mmol/L), CFB, wk36 (N=4, N=2) | -0.3 (0.7) | 0.1 (0.5)
  Triglyceride (mmol/L), CFB, EoT (N=67, N=73) | 0.1 (0.6) | 0.1 (0.6)
  Glucose (mmol/L), CFB, day1 (N=76, N=75) | -0.1 (1.3) | 0.2 (0.9)
  Glucose (mmol/L), CFB, wk2 (N=75, N=78) | -0.1 (1.3) | 0.1 (1.0)
  Glucose (mmol/L), CFB, wk4 (N=74, N=77) | -0.2 (1.3) | 0.1 (0.9)
  Glucose (mmol/L), CFB, wk8 (N=74, N=76) | -0.1 (1.3) | 0.1 (0.9)
  Glucose (mmol/L), CFB, wk12 (N=73, N=76) | -0.3 (1.1) | -0.1 (1.0)
  Glucose (mmol/L), CFB, wk18 (N=67, N=70) | -0.4 (1.2) | -0.1 (0.7)
  Glucose (mmol/L), CFB, wk24 (N=12, N=4) | -0.7 (1.3) | -0.4 (0.7)
  Glucose (mmol/L), CFB, wk28 (N=5, N=3) | -0.4 (1.1) | 0.1 (0.7)
  Glucose (mmol/L), CFB, wk36 (N=4, N=2) | -0.1 (0.7) | -0.1 (0.4)
  Glucose (mmol/L), CFB, EoT (N=66, N=71) | -0.4 (1.2) | -0.1 (1.3)

15. Secondary Outcome: Laboratory Test Value Changes Over Time for Selected Lab Test Parameters (5)
Description: Change from baseline (CFB) in AST/GOT, ALT/GPT, Alka. phosphatase, GGT, Creatine kinase, Lipase, and Amylase.
Time Frame: baseline and 48 weeks
Population: TS
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Faldaprevir 120mg (12 Weeks) | Faldaprevir 120mg (24 Weeks)
Number analyzed (Participants) | 81 | 79
U/L
  AST/GOT (U/L), CFB, Day 1(N=74, N=75) | 0 (28) | -5 (29)
  AST/GOT (U/L), CFB, wk2 (N=75, N=78) | -24 (30) | -29 (43)
  AST/GOT (U/L), CFB, wk4 (N=74, N=76) | -25 (31) | -29 (49)
  AST/GOT (U/L), CFB, wk8 (N=74, N=76) | -22 (36) | -27 (47)
  AST/GOT (U/L), CFB, wk12 (N=74, N=76) | -24 (29) | -27 (44)
  AST/GOT (U/L), CFB, wk18 (N=67, N=70) | -25 (33) | -30 (50)
  AST/GOT (U/L), CFB, wk24 (N=12, N=4) | -23 (60) | -10 (15)
  AST/GOT (U/L), CFB, wk28 (N=5, N=3) | -20 (27) | -16 (24)
  AST/GOT (U/L), CFB, wk36 (N=4, N=2) | -21 (40) | 11 (4)
  AST/GOT (U/L), CFB, EoT (N=66, N=71) | -25 (41) | -27 (49)
  ALT/GPT (U/L), CFB, day1 (N=76, N=75) | 1 (24) | -2 (22)
  ALT/GPT (U/L), CFB, wk2 (N=75, N=78) | -37 (36) | -34 (40)
  ALT/GPT (U/L), CFB, wk4 (N=74, N=77) | -37 (40) | -34 (50)
  ALT/GPT (U/L), CFB, wk8 (N=74, N=76) | -36 (43) | -35 (49)
  ALT/GPT (U/L), CFB, wk12 (N=74, N=76) | -37 (36) | -36 (48)
  ALT/GPT (U/L), CFB, wk18 (N=67, N=70) | -41 (40) | -42 (52)
  ALT/GPT (U/L), CFB, wk24 (N=12, N=4) | -40 (50) | -24 (22)
  ALT/GPT (U/L), CFB, wk28 (N=5, N=3) | -45 (38) | -22 (15)
  ALT/GPT (U/L), CFB, wk36 (N=4, N=2) | -47 (46) | -6 (4)
  ALT/GPT (U/L), CFB, EoT (N=66, N=71) | -42 (42) | -42 (45)
  Alka. phosphatase (U/L), CFB, day1 (n=77, N=75) | 1 (11) | 1 (13)
  Alka. phosphatase (U/L), CFB, wk2 (n=76, N=78) | 5 (10) | 7 (11)
  Alka. phosphatase (U/L), CFB, wk4 (n=76, N=77) | 7 (13) | 10 (13)
  Alka. phosphatase (U/L), CFB, wk8 (n=75, N=76) | 7 (13) | 9 (15)
  Alka. phosphatase (U/L), CFB, wk12 (n=75, N=76) | 5 (14) | 6 (14)
  Alka. phosphatase (U/L), CFB, wk18 (n=68, N=70) | -2 (20) | 5 (14)
  Alka. phosphatase (U/L), CFB, wk24 (n=12, N=4) | -14 (24) | 13 (13)
  Alka. phosphatase (U/L), CFB, wk28 (n=5, N=3) | -2 (14) | 15 (3)
  Alka. phosphatase (U/L), CFB, wk36 (n=4, N=2) | -5 (16) | 18 (4)
  Alka. phosphatase (U/L), CFB, EoT (n=67, N=73) | 1 (22) | 5 (16)
  GGT (U/L), CFB, day1 (N=77, N=75) | -5 (39) | -5 (88)
  GGT (U/L), CFB, wk2 (N=76, N=78) | -34 (71) | -38 (117)
  GGT (U/L), CFB, wk4 (N=76, N=77) | -59 (86) | -60 (135)
  GGT (U/L), CFB, wk8 (N=75, N=76) | -76 (96) | -70 (143)
  GGT (U/L), CFB, wk12 (N=75, N=76) | -71 (103) | -69 (150)
  GGT (U/L), CFB, wk18 (N=68, N=70) | -62 (105) | -64 (146)
  GGT (U/L), CFB, wk24 (N=12, N=4) | -118 (200) | -131 (50)
  GGT (U/L), CFB, wk28 (N=5, N=3) | -52 (126) | -113 (42)
  GGT (U/L), CFB, wk36 (N=4, N=2) | -23 (132) | -14 (73)
  GGT (U/L), CFB, EoT (N=67, N=73) | -39 (106) | -59 (148)
  Creatine kinase (U/L), CFB, day1 (N=76, N=75) | -2 (140) | 30 (308)
  Creatine kinase (U/L), CFB, wk2 (N=75, N=78) | -59 (158) | -41 (118)
  Creatine kinase (U/L), CFB, wk4 (N=74, N=77) | -69 (173) | -62 (134)
  Creatine kinase (U/L), CFB, wk8 (N=74, N=76) | -92 (176) | -75 (131)
  Creatine kinase (U/L), CFB, wk12 (N=74, N=75) | -98 (186) | -84 (132)
  Creatine kinase (U/L), CFB, wk18 (N=67, N=70) | -93 (202) | -60 (216)
  Creatine kinase (U/L), CFB, wk24 (N=12, N=4) | -69 (78) | -42 (30)
  Creatine kinase (U/L), CFB, wk28 (N=5, N=3) | -48 (75) | -32 (26)
  Creatine kinase (U/L), CFB, wk36 (N=4, N=2) | -68 (83) | -37 (22)
  Creatine kinase (U/L), CFB, EoT (N=66, N=71) | -89 (187) | -21 (331)
  Lipase (U/L). CFB, day1 (N=77, N=75) | -2 (52) | 26 (239)
  Lipase (U/L). CFB, wk2 (N=76, N=78) | 5 (65) | 9 (30)
  Lipase (U/L). CFB, wk4 (N=76, N=76) | -1 (52) | 6 (36)
  Lipase (U/L). CFB, wk8 (N=75, N=76) | -11 (69) | 2 (57)
  Lipase (U/L). CFB, wk12 (N=75, N=75) | -12 (70) | 4 (90)
  Lipase (U/L). CFB, wk18 (N=68, N=70) | -13 (64) | -4 (32)
  Lipase (U/L). CFB, wk24 (N=12, N=4) | 2 (31) | -17 (22)
  Lipase (U/L). CFB, wk28 (N=5, N=3) | -1 (13) | 0 (11)
  Lipase (U/L). CFB, wk36 (N=4, N=2) | -4 (12) | -15 (0)
  Lipase (U/L). CFB, EoT (N=67, N=73) | -6 (82) | -5 (27)
  Amylase (U/L), CFB, day1 (N=77, N=75) | 1 (26) | 7 (68)
  Amylase (U/L), CFB, wk2 (N=76, N=78) | 5 (41) | 3 (23)
  Amylase (U/L), CFB, wk4 (N=76, N=77) | 2 (30) | 5 (27)
  Amylase (U/L), CFB, wk8 (N=75, N=76) | -5 (33) | -2 (29)
  Amylase (U/L), CFB, wk12 (N=75, N=75) | -10 (33) | -4 (33)
  Amylase (U/L), CFB, wk18 (N=68, N=70) | -7 (34) | -7 (28)
  Amylase (U/L), CFB, wk24 (N=12, N=4) | -14 (35) | -16 (23)
  Amylase (U/L), CFB, wk28 (N=5, N=3) | -21 (34) | -8 (7)
  Amylase (U/L), CFB, wk36 (N=4, N=2) | -35 (24) | -19 (9)
  Amylase (U/L), CFB, EoT (N=67, N=73) | 0 (37) | -4 (27)

16. Secondary Outcome: Laboratory Test Value Changes Over Time for Selected Lab Test Parameters (6)
Description: Change from baseline (CFB) in PT-INR (ratio).
Time Frame: baseline and 48 weeks
Population: TS
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Faldaprevir 120mg (12 Weeks) | Faldaprevir 120mg (24 Weeks)
Number analyzed (Participants) | 81 | 79
ratio
  PT-INR (ratio), CFB, Day 1(N=77, N=72) | 0.0 (0.2) | 0.0 (0.1)
  PT-INR (ratio), CFB, wk2 (N=76, N=78) | 0.0 (0.1) | 0.0 (0.1)
  PT-INR (ratio), CFB, wk4(N=74, N=76) | 0.0 (0.1) | 0.0 (0.1)
  PT-INR (ratio), CFB, wk8(N=73, N=75) | 0.0 (0.1) | 0.0 (0.1)
  PT-INR (ratio), CFB, wk12(N=74, N=72) | 0.0 (0.1) | 0.0 (0.1)
  PT-INR (ratio), CFB, wk18(N=69, N=70) | 0.0 (0.1) | 0.0 (0.1)
  PT-INR (ratio), CFB, wk24(N=12, N=4) | 0.0 (0.1) | 0.1 (0.1)
  PT-INR (ratio), CFB, wk28(N=5, N=3) | -0.1 (0.1) | 0.0 (0.1)
  PT-INR (ratio), CFB, wk36(N=4, N=2) | 0.0 (0.1) | -0.1 (0.1)
  PT-INR (ratio), CFB, EoT(N=68, N=73) | 0.0 (0.1) | 0.0 (0.1)

ADVERSE EVENTS:
Time Frame: up to 24 weeks + 30 days washout.
Description: One patient, randomised to the 12 week treatment, received PegIFN/RBV during the lead-in phase but never started treatment with Faldaprevir and therefore is not included in the adverse event summary.
Groups:
- Faldaprevir 120 mg (12 Weeks): Patients received Faldaprevir (BI201335) 120 mg soft gelatine capsule once daily combined with PegIFN/RBV (Pegylated interferon alpha-2a solution for injection/Ribavirin tablet) for 12 weeks, with a 3 days lead-in phase of PegIFN/RBV (i.e. initiation of Faldaprevir (BI201335) 3 days after first administration of PegIFN/RBV), followed by PegIFN/RBV for additional 12 weeks.
- Faldaprevir 120 mg (24 Weeks): Patients received Faldaprevir (BI201335) 120 mg soft gelatine capsule once daily combined with PegIFN/RBV (Pegylated interferon alpha-2a solution for injection/Ribavirin tablet) for 24 weeks, with a 3 days lead-in phase of PegIFN/RBV (i.e. initiation of Faldaprevir (BI201335) 3 days after first administration of PegIFN/RBV).
Arm/Group | Faldaprevir 120 mg (12 Weeks) | Faldaprevir 120 mg (24 Weeks)
Serious Adverse Events (participants affected / at risk) | 3/80 | 3/79
Other Adverse Events (participants affected / at risk) | 73/80 | 68/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Faldaprevir 120 mg (12 Weeks) (N=80) | Faldaprevir 120 mg (24 Weeks) (N=79)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Faldaprevir 120 mg (12 Weeks) (N=80) | Faldaprevir 120 mg (24 Weeks) (N=79)
Anaemia (Blood and lymphatic system disorders) | 6 | 13
Neutropenia (Blood and lymphatic system disorders) | 3 | 7
Vertigo (Ear and labyrinth disorders) | 5 | 0
Dry eye (Eye disorders) | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 5
Abdominal pain upper (Gastrointestinal disorders) | 4 | 4
Constipation (Gastrointestinal disorders) | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 15
Dry mouth (Gastrointestinal disorders) | 7 | 2
Nausea (Gastrointestinal disorders) | 27 | 17
Vomiting (Gastrointestinal disorders) | 11 | 7
Asthenia (General disorders) | 18 | 13
Fatigue (General disorders) | 17 | 13
Influenza like illness (General disorders) | 5 | 7
Irritability (General disorders) | 4 | 7
Jaundice (Hepatobiliary disorders) | 3 | 4
Bronchitis (Infections and infestations) | 2 | 5
Decreased appetite (Metabolism and nutrition disorders) | 14 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Disturbance in attention (Nervous system disorders) | 3 | 6
Dizziness (Nervous system disorders) | 4 | 4
Headache (Nervous system disorders) | 14 | 18
Anxiety (Psychiatric disorders) | 3 | 7
Depression (Psychiatric disorders) | 7 | 13
Insomnia (Psychiatric disorders) | 9 | 15
Sleep disorder (Psychiatric disorders) | 3 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 12 | 16
Eczema (Skin and subcutaneous tissue disorders) | 3 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 24 | 26
Rash (Skin and subcutaneous tissue disorders) | 18 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.